CLINICAL TRIAL: NCT02669303
Title: Comparing Subacromial Injection of Platelet-rich Plasma Versus Methylprednisolone in the Treatment of Shoulder Subacromial Impingement Syndrome
Brief Title: Platelet-rich Plasma (PRP) Injection for Treating Shoulder Subacromial Impingement Syndrome
Acronym: ShIP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment rate and high rate of loss-to-followup
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Muhyeddine Al-Taki, Assistant Professor of Clinical Surgery, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SUR.MA.134
Record Dates: First submitted 2015-10-15; First posted 2016-02-01 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Subacromial injection; methylprednisolone; treatment; Platelet-rich plasma
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- platelet-rich plasma group (Experimental): Autologous platelet-rich plasma subacromial injection
  Interventions: Drug: platelet-rich plasma group
- Methylprednisolone group (Active Comparator): Methylprednisolone subacromial injection
  Interventions: Drug: Methylprednisolone group

INTERVENTIONS:
Drug: platelet-rich plasma group — Once randomized to platelet-rich plasma arm, the study subject will have 30cc of blood drawn and centrifuged using the "Recover(TM) Platelet Separation Kit" (Biomet Biologics, Warsaw, Indiana, USA). The extracted platelet-rich plasma part will be re-injected into the subacromial space of the subject's affected shoulder.
  Other Names: autologous platelet-rich plasma; PRP
  Arms: platelet-rich plasma group
Drug: Methylprednisolone group — Once randomized to Methylprednisolone arm, the study subject will have an injection with 2ml of Methylprednisolone (40mg/ml methylprednisolone acetate injectable suspension) (Pharmacia Upjohn, Kalamazoo, Michigan, USA) with 2ml of lidocaine hydrochloride 2% (Hameln Pharmaceuticals Ltd, Gloucester, UK) into the subacromial space of their affected shoulder.
  Other Names: methylprednisolone acetate
  Arms: Methylprednisolone group

SUMMARY:
The purpose of this study is to determine whether injection of platelet-rich plasma derived from patient's blood is effective in treatment of shoulder subacromial impingement syndrome as compared to the current protocol of methylprednisolone injection.

DETAILED DESCRIPTION:
Patients presenting with shoulder pain to the study location will be screened by the principal investigator. Once diagnosed clinically with shoulder subacromial impingement syndrome, they will be invited to join the study. They will be invited to separate academic office to be explained about the study, its voluntary and confidential basis as per our Institutional Review Board (IRB) approved protocols.

After signing informed consent form and recruitment, they will be assigned randomly to one of the study arms through software-generated sequential allocation packaged in an opaque envelope. All involved except the principal investigator and patient are blinded.

There are two groups/arms in the study. The experimental arm will include subacromial injection of study subjects with autologous platelet-rich plasma; wheres subjects in the other study arm will be injected with methylprednisolone.

The outcome will be assessed through three scores. The study subjects will be asked to complete Oxford Shoulder Score questionnaire and health-related quality of life SF-36 questionnaire and Constant-Murley score will be measured through physician-based assessment done by the residents involved in the study. This will be done during the baseline visit before injection and repeated at 2, 6, 12 weeks and 6 months follow-up visits.

Also any adverse effects of both treatment arms will be monitored and reported as appropriate.

The investigators hypothesize that injecting platelet-rich plasma into the subacromial space of patients with subacromial impingement will result in decreased pain and increased function at 6 months follow-up (assessed by Constant-Murley Score, Oxford Shoulder Score, and Short Form-36 (SF-36) questionnaire) as compared to patients injected with methylprednisolone.

ELIGIBILITY:
Inclusion Criteria:

* Any adult male or female between 18 and 65 years of age, inclusive, with clinical diagnosis of shoulder subacromial impingement

Exclusion Criteria:

* Age below 18 or above 65 years
* History of prior shoulder injections or surgery
* History of fracture of the acromion, clavicle, scapula, or proximal humerus
* Known allergy to corticosteroids
* Known allergy to lidocaine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Constant-Murley Total Score | 6 months post-injection
  The sum of scores from different domains of Constant-Murley Questionnaire

SECONDARY OUTCOMES:
Constant-Murley Pain Score | 6 months post-injection
  Pain score derived from Pain domain of Constant-Murley Questionnaire
Constant-Murley Function score | 6 months post-injection
  Function score derived from function domain of Constant-Murley Questionnaire
Constant-Murley ROM score | 6 months post-injection
  Range of motion assessment score derived from range of motion domain of Constant-Murley Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Muhyeddine Al-Taki, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gosens T, Peerbooms JC, van Laar W, den Oudsten BL. Ongoing positive effect of platelet-rich plasma versus corticosteroid injection in lateral epicondylitis: a double-blind randomized controlled trial with 2-year follow-up. Am J Sports Med. 2011 Jun;39(6):1200-8. doi: 10.1177/0363546510397173. Epub 2011 Mar 21. PMID 21422467
- [Background] Anitua E, Andia I, Sanchez M, Azofra J, del Mar Zalduendo M, de la Fuente M, Nurden P, Nurden AT. Autologous preparations rich in growth factors promote proliferation and induce VEGF and HGF production by human tendon cells in culture. J Orthop Res. 2005 Mar;23(2):281-6. doi: 10.1016/j.orthres.2004.08.015. PMID 15779147
- [Background] Karthikeyan S, Kwong HT, Upadhyay PK, Parsons N, Drew SJ, Griffin D. A double-blind randomised controlled study comparing subacromial injection of tenoxicam or methylprednisolone in patients with subacromial impingement. J Bone Joint Surg Br. 2010 Jan;92(1):77-82. doi: 10.1302/0301-620X.92B1.22137. PMID 20044683